CLINICAL TRIAL: NCT05689788
Title: Effect of High-intensity Laser Therapy in Patients With Chronic Nonspecific Neck Pain. Randomized Clinical Trial
Brief Title: High-intensity Laser Therapy for Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Principal Investigator, Hernán Andrés de la Barra Ortiz, Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26122022
Record Dates: First submitted 2022-12-26; First posted 2023-01-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Non-specific Chronic Neck Pain
Keywords: Lasers; Laser therapy; Chronic pain; Neck pain; Physical Therapy Modalities; Clinical trial
MeSH Terms: conditions — Chronic Pain; Neck Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT + stretching exercise (Experimental): High-intensity laser therapy (HILT) will be applied with the punctual technique on the 6 bilateral points of the cervical region and shoulder girdle, to be followed by a sweep technique on both trapezius muscles (upper portions). The parameters proposed by Dundar et al. will be used: an average power of 3 W, 60 J per point (360 J), and 500 J for manual scanning (1000 J). For the application of laser therapy, the 12 W BTL-6000 equipment that emits at 1064 nm wavelengths will be used. Laser therapy will be applied with the participant in the prone position.The treatment will be complemented with passive static stretching for the upper trapezius, levator scapulae, and scalene muscles (bilaterally) in three series. Each series will last 30 seconds, followed by a 30-second rest interval. The exercises will be carried out with the participant in a seated position in a chair with a backrest.
  Interventions: Device: High-intensity laser therapy; Procedure: Stretching exercise
- Sham HILT + stretching exercise (Sham Comparator): The group will receive a sham treatment of high-intensity laser therapy (HILT). The treatment will be complemented with passive static stretching for the upper trapezius, levator scapulae, and scalene muscles (bilaterally) in three series. Each series will last 30 seconds, followed by a 30-second rest interval. The exercises will be carried out with the participant in a seated position in a chair with a backrest.
  Interventions: Procedure: Stretching exercise; Device: Sham High-intensity laser therapy

INTERVENTIONS:
Device: High-intensity laser therapy — punctual technique on the 6 bilateral points of the cervical region and shoulder girdle, to be followed by a sweep technique on both trapezius muscles (upper portions). The parameters proposed by Dundar et al. will be used: an average power of 3 W, 60 J per point (360 J), and 500 J for manual scanning (1000 J). For the application of laser therapy, the 12 W BTL-6000 equipment that emits at 1064 nm wavelengths will be used.
  Arms: HILT + stretching exercise
Procedure: Stretching exercise — Three sets of bilateral passive static stretching will be performed for the upper trapezius, levator scapulae, and scalene muscles. Each series will last 30 seconds, followed by a 30-second rest interval. The exercises will be carried out with the participant in a seated position in a chair with a backrest.
Device: Sham High-intensity laser therapy — Intervention in which the therapist performs a HILT simulation application, performing all of the steps and movements for an administration without actually receiving the treatment.
  Arms: Sham HILT + stretching exercise

SUMMARY:
Chronic nonspecific neck pain is a common musculoskeletal disorder recognized for its high rates of disability and economic losses, ranking second in musculoskeletal conditions after low back pain. There are several effective physical therapy interventions to treat chronic nonspecific neck pain, such as laser therapy. High-intensity laser therapy (HILT) is a recent treatment proposed to reduce musculoskeletal pain; however, there are few studies that prove its effects in reducing neck pain.

The aim of this randomized clinical trial is to evaluate the effect of high-intensity laser therapy on pain intensity in patients with chronic nonspecific neck pain.

The research will be carried out in the laboratory of physical agents at the Andrés Bello University, Campus Casona de las Condes. Participants will be employers and volunteer students with non-specific chronic neck pain. Participants will be randomized and allocated into 2 study groups: group 1 (HILT and stretching exercises) and group 2 (simulated HILT and stretching exercises). Treatments will be performed twice a week for 4 weeks with 3 assessments: before treatment, at the end of treatment, and 12 weeks after treatment (follow-up). The main results will be the differences in pain pressure threshold (ΔPPT), intensity of pain at rest (ΔRPI) and intensity of pain on movement (ΔMPI). Secondary outcome measures, on the other hand, will include differences in cervical spine range (ΔCROM) and cervical disability (ΔND).

DETAILED DESCRIPTION:
Material and Methods

Type of study: Experimental, randomized clinical trial (RCT).

1. Study population:

   For the study, students and employees of Andrés Bello University will be considered participants.
2. Randomization and sample:

   Participants will be evaluated according to the selection criteria through a survey with closed questions and a clinical examination that will determine the presence or absence of chronic non-specific neck pain. Participants will be divided into two study groups through a simple randomization process: group 1 (HILT) and group 2 (sham HILT). The randomization of the sample will be carried out by the study director using the simple random sampling process through the research randomizer program, who will be the only one who knows the results. All groups will receive a treatment with an exercise plan that includes passive static stretching of the upper trapezius, levator scapulae, and scalenes muscles (three sets of 30 seconds for each group bilaterally). Participants will be scheduled twice a week for four weeks to carry out the assigned treatment.

   The sample size was determined with the G-Power program using a power of 0.80 (1-β), a reliability of 95%, an error of 5% (α) and an effect size of 0.6 (d- Cohen) with reference to previous studies that determined differences in mean pain intensity between experimental and control groups after HILT treatment with effect sizes of 0.53. Based on the above, the sample size is 72 subjects, with at least 36 subjects per group.
3. Procedures The outcomes to be measured will be: pain pressure threshold (PPT), resting pain intensity (RPI), movement pain intensity (MPI), cervical range of motion (CROM), and cervical disability (ND).

   Pain pressure threshold (PPT) will be evaluated with pressure algometry at six bilateral points established for the cervical region and shoulders, pain intensity at rest and on movement with VAS (RPI and MPI), cervical ROM with an inclinometer (CROM system), and cervical disability (ND) through the cervical disability index (NDI). The evaluations will be carried out by 2 independent evaluators: evaluator 1, PPT with algometry and PI with VAS (RPI and MPI); and evaluator 2, CROM with cervical inclinometry and ND with the cervical disability index. The PPT values will be evaluated in kg/cm2, the MPI will be evaluated in millimeters, the CROM will be evaluated in degrees for all movements of the cervical spine, and the ND will be evaluated as a percentage of disability. Values for the outcome measures of interest will be tabulated in an Excel® spreadsheet by each rater.

   The evaluations will be carried out during the study in three instances (T0-T1), including a later follow-up evaluation (T3): pretreatment (T0: baseline), end of treatment at 8 weeks (T1), and twelve weeks (T3: follow-up). The participants will be summoned twice a week to carry out their corresponding treatments. On the other hand, cervical disability will be evaluated using the Spanich version of Neck Disability Index (NDI), obtaining the percentage of disability for each of the evaluation instances. Moreover, the NDI will be applied as a self-report before and after the treatment sessions (T0 and T2).

   Once the study is over, the differences in cervical range of motion (ΔCFROM), pain pressure threshold (ΔPPT), pain intensity at rest (ΔRPI), pain intensity at movement (ΔMPI) and cervical disability (ΔNDI) between the evaluation sessions will be evaluated.
4. Variables

   4.1 Conceptual definition of the variables
   * Painful pressure threshold (PPT): the magnitude of pressure described as painful by the participant when performing the six-point algometry test in the cervical and shoulder regions: 2 cm lateral to the spinous processes of C2, C5, T4, and T8, midpoint of the upper portion of the trapezius muscle belly (between the spinous process of C7 and the acromion), and levator scapula muscle (2 cm superior to the superior angle of the scapula).
   * Pain intensity at rest (RPI): the magnitude of neck pain reported by participants when they are at rest.
   * Movement pain intensity (MPI): magnitude of pain reported by the participants when performing movements of the cervical spine in flexion, extension, inclination, and right and left rotation.
   * Cervical range of motion (CROM): range of motion of the head relative to the trunk for flexion, extension, right tilt, left tilt, right rotation, and left rotation movements.
   * Neck disability (ND): lack or limitation of the functionality of the cervical region due to pain that makes it impossible or difficult to carry out normal activities of daily living.
   * High Intensity Laser Therapy (HILT): laser application with powers greater than 500 milliwatts (mW) at the algometry assessment points and upper trapezius muscle belly.
   * Stretching exercise (SE): Bilateral passive static stretching for the upper trapezius, levator scapulae, and scalenes muscles.

   4.2 Operational definition of variables.
   * Painful Pressure Threshold (PPT): The painful pressure threshold (PPT) will be quantified by pressure algometry, recording the sum of the values in kg/cm2 of pressure for the six bilateral points established to perform the measurement. Three measurements will be made for each point with an interval of 30 seconds, recording the average of the three as the final value. For the evaluation, the Baseline® brand pressure algometer will be used. The PPT exam will be performed by placing the participant in a prone position. The intra-rater reliability for the PPT measurement will be determined with the intra-class coefficient by assessing the PPT at the upper trapezius muscle belly point in 13 healthy volunteers not involved in the study with a 48-h interval between assessments.
   * Pain intensity at rest (RPI): Pain intensity will be assessed using a visual analogue scale (VAS) (ICC = 0.97 (CI 95% 0.96, 0.98) [30]. The RPI The MPI exam will be carried out by the participant in a seated position, keeping the back straight and supported on a backrest.
   * Movement pain intensity (MPI): Pain intensity will be assessed through the visual analogue scale (VAS) for movements of flexion, extension, inclination, and cervical rotation. The MPI value will correspond to the sum of the VAS score for all cervical movements. The MPI exam will be carried out by the participant in a seated position, keeping the back straight and supported on a backrest.
   * Cervical range of motion (CROM): The range of cervical motion will be evaluated through an inclinometer, recording the degrees of movement for the movements of flexion, extension, right tilt, left tilt, right rotation, and left rotation. To measure the range of motion, the CROM device will be used (inter-evaluator reliability: Extension ICC = 0.98 (CI 95% 0.95, 0.99); Flexion ICC = 0.89 (CI 95% 0.73,0.96); Left rotation ICC = 0.95 (CI 95 % 0.87, 0.98); Rotation right ICC = 0.92 (CI 95% 0.80, 0.97); Tilt left ICC = 0.97 (CI 95% 0.91, 0.99); Tilt right ICC = 0.97 (CI 95% 0.93, 0.99). The CROM examination will be performed while seated with a straight back and supported by the chair's back.
   * Neck disability (ND): Neck disability will be assessed through the Neck Disability Index (NDI), an instrument consisting of 10 sections with questions related to symptoms and life activities that may be limited by neck pain and that has been validated for the Spanish language. Each section consists of questions scored from 0-5, with greater disability being associated with a higher score (NDI; inter-rater reliability: ICC = 0.93 (95% CI 0.86, 0.97).
   * High-Intensity Laser Therapy (HILT): High intensity laser therapy (HILT) will be applied with the punctual technique on the 6 bilateral points of the cervical region and shoulder girdle, to be followed by a sweep technique on both trapezius muscles. Dundar et al. propose the following parameters: a 3 watt average power, 60 joules per point (360 joules), and 500 joules for manual scanning (1000 joules). For the application of laser therapy, the 12 W BTL-6000 equipment that emits at 1064 nm wavelengths will be used. Laser therapy will be applied with the participant in the prone position.
   * Stretching exercise (SE): Three sets of bilateral passive static stretching will be performed for the upper trapezius, levator scapulae, and scalene muscles. Each series will last 30 seconds, followed by a rest interval of 30 seconds. The exercises will be carried out with the participant in a seated position in a chair with a backrest.

   4.3 Variable type definition
   * Painful Pressure Threshold (PPT): dependent, quantitative, continuous variable.
   * Pain intensity on movement (MPI): dependent, quantitative, discrete variable.
   * Cervical range of motion (CROM): dependent, quantitative, discrete variable.
   * Cervical disability (ND): dependent, quantitative, continuous variable.
   * High Intensity Laser Therapy (HILT): independent, quantitative, continuous variable.
   * Stretching exercise (EE): independent, quantitative, discrete variable.
5. Study phases Three phases have been designated for the investigation: Sampling phase, Evaluation phase and Intervention phase.

   The sampling phase will consist of applying the selection survey to potential participants. Participants will be chosen according to the selection criteria through a survey that will determine the presence of non-specific chronic neck pain (CNCP). The survey will be conducted online using a Microsoft Office® form. The selected participants will be divided into two study groups through a simple randomization process (research randomizer, https://www.randomizer.org/): group 1 (HILT + stretching exercise) and group 2 (sham HILT + stretching exercise). The randomization of the sample will be carried out by the study director, using the simple random sampling process through the research randomizer program, who will be the only one who knows the results. Participants will meet twice a week for four weeks to carry out the assigned treatment.

   The evaluation phase will consist of measuring the outcomes of interest. Pain pressure threshold (PPT) will be evaluated with pressure algometry at six established bilateral points, pain intensity at rest and on movement with VAS (RPI and MPI), cervical ROM with an inclinometer (CROM system), and the neck disability (ND) through the spanich version of Neck Disability Index. The evaluations of the interest outcome measures will be carried out in three instances; pretreatment (T0: baseline), the fourth week (T2: 8th session, end of treatment), and week 20 (T3: 12 weeks post-treatment or follow-up). The differences in pain pressure threshold (ΔPPT), pain intensity at rest (ΔRPI) and pain intensity on movement (ΔMPI) will be considered the main outcome measures. Alternatively, secondary outcome measures will include differences in cervical spine range (ΔCROM) and cervical disability (ΔND).

   The intervention phase will include eight treatment sessions held twice a week to carry out their corresponding treatments (4 weeks total). The sample will be treated in two study groups: the HILT group and the sham HILT group. All groups will receive, as a base treatment, a passive static cervical stretching therapeutic exercise plan focused on the upper trapezius, levator scapulae, and scalene muscles of three series for 30 seconds. The interventions will be carried out by two independent, trained therapists.The participants will be summoned twice a week to carry out their corresponding treatments.
6. Statistic analysis

The descriptive statistics for the primary variables ΔPPT, ΔRPI, ΔMPI ΔCROM, and ΔND will use as analysis measures, means and standard deviation (x, SD), or median and interquartile range (mean, IQR), depending on the distribution of the data (test of normality of Kolmogorov-Smirnov). This will make it possible to build the table with the demographic data of the participants by group (Table 1 of the work). According to the data normality analysis, frequencies and means or medians will be used for the secondary variables sex and body mass index (BMI).For inferential statistical analysis of the outcome measures of interest obtained between assessments, the Kolmogorov-Smirnov normality test will be used to determine their distribution. According to the results, parametric or non-parametric tests will be selected: the T-test for independent samples if the data is normally distributed or the U-Mann Whitney test if the variables are not normally distributed. For statistical analysis, the IBM SPSS (Statistical Package for the Social Sciences) v26 program will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old.
* Both sexes (men and women)
* Non-specific, chronic neck pain, defined as pain or discomfort in the cervical region between the superior nuchal line and the spinous process of T1 or the shoulder girdle, with the following criteria: neck pain in the last 3 months or more; a questionnaire score of cervical disability (NDI) equal to or greater than 5; and cervical pain of 3 or greater on the numerical pain scale (NPRS).

Exclusion Criteria:

* Neck or shoulder musculoskeletal injuries in the last 3 months (fractures, sprains, tendinopathies, dislocations, or muscle tears).
* Osteosynthesis materials close to the shoulders, neck, or surrounding areas.
* Wounds or skin changes in the shoulder and/or neck region (such as psoriasis, scars, or burns).
* Analgesic, anti-inflammatory, or muscle relaxant drugs for permanent use.
* Neurological alterations such as paresthesia, loss of sensation (partial or complete), decrease in strength, or color changes in the neck, arms, forearms, or hands.
* Diagnosed photosensitivity.
* Presence of solar urticaria or adverse reactions to sunlight.
* The presence of dermatomyositis, systemic lupus erythematosus, hepatic porphyria, cutaneous carcinoid syndrome, or pellagra.
* Cancer or tumors of some type have been diagnosed in the last 5 years.
* Epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Pain pressure thereshold (PPT) | Baseline, 4 weeks (8 sessions) and 12 weeks (follow-up)
  Pain pressure threshold differences evaluated with algometry at six neck and shoulder locations: 2 cm lateral to the spinous processes of C2, C5, T4, and T8, midpoint of the upper trapezius muscle belly (between the spinous process of C7 and the acromion), and the levator scapula muscle (2 cm superior to the superior angle of the scapula).
Pain intensity at rest (RPI) | Baseline, 4 weeks (8 sessions) and 12 weeks (follow-up)
  Magnitude of neck pain reported by participants at rest evaluated with visual anologue scale (VAS)
Pain intensity at movement (MPI) | Baseline and 4 weeks (8 sessions)
  Magnitude of pain reported by the participants when performing movements of the cervical spine in flexion, extension, inclination, and right and left rotation evaluated with visual anologue scale (VAS).

SECONDARY OUTCOMES:
Cervical range of motion (CROM) | Baseline and 4 weeks (8 sessions)
  Range of motion of the head relative to the trunk in flexion, extension, right tilt, left tilt, right rotation, and left rotation movements evalluated with goniometry (cervical ROM device).
Neck disability (ND) | Baseline and 4 weeks (8 sessions)
  Lack or limitation of the functionality of the cervical region due to pain makes it impossible or difficult to carry out normal activities of daily living evaluated with the Neck Disability Index (NDI)

CONTACTS AND LOCATIONS:
Overall Officials: Hernán de la Barra Ortiz, MSc, Principal Investigator — Universidad Andrés Bello
Locations (2):
- Chile (2):
  - Universidad Andrés Bello, Santiago, Las Condes
  - Hernán Andrés de la Barra, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Fandim JV, Nitzsche R, Michaleff ZA, Pena Costa LO, Saragiotto B. The contemporary management of neck pain in adults. Pain Manag. 2021 Jan;11(1):75-87. doi: 10.2217/pmt-2020-0046. Epub 2020 Nov 25. PMID 33234017
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] Peron R, Rampazo EP, Liebano RE. Traditional acupuncture and laser acupuncture in chronic nonspecific neck pain: study protocol for a randomized controlled trial. Trials. 2022 May 16;23(1):408. doi: 10.1186/s13063-022-06349-y. PMID 35578302
- [Background] Alayat MS, Mohamed AA, Helal OF, Khaled OA. Efficacy of high-intensity laser therapy in the treatment of chronic neck pain: a randomized double-blind placebo-control trial. Lasers Med Sci. 2016 May;31(4):687-94. doi: 10.1007/s10103-016-1910-2. Epub 2016 Feb 25. PMID 26914684
- [Background] Matre D, Knardahl S. 'Central sensitization' in chronic neck/shoulder pain. Scand J Pain. 2012 Oct 1;3(4):230-235. doi: 10.1016/j.sjpain.2012.04.003. PMID 29913871
- [Background] Diwan S, Manchikanti L, Benyamin RM, Bryce DA, Geffert S, Hameed H, Sharma ML, Abdi S, Falco FJ. Effectiveness of cervical epidural injections in the management of chronic neck and upper extremity pain. Pain Physician. 2012 Jul-Aug;15(4):E405-34. PMID 22828692
- [Background] Cotler HB, Chow RT, Hamblin MR, Carroll J. The Use of Low Level Laser Therapy (LLLT) For Musculoskeletal Pain. MOJ Orthop Rheumatol. 2015;2(5):00068. doi: 10.15406/mojor.2015.02.00068. Epub 2015 Jun 9. PMID 26858986
- [Background] Hadis MA, Zainal SA, Holder MJ, Carroll JD, Cooper PR, Milward MR, Palin WM. The dark art of light measurement: accurate radiometry for low-level light therapy. Lasers Med Sci. 2016 May;31(4):789-809. doi: 10.1007/s10103-016-1914-y. Epub 2016 Mar 10. PMID 26964800
- [Background] Khalkhal E, Razzaghi M, Rostami-Nejad M, Rezaei-Tavirani M, Heidari Beigvand H, Rezaei Tavirani M. Evaluation of Laser Effects on the Human Body After Laser Therapy. J Lasers Med Sci. 2020 Winter;11(1):91-97. doi: 10.15171/jlms.2020.15. Epub 2020 Jan 18. PMID 32099633
- [Background] Stewart N, Lim AC, Lowe PM, Goodman G. Lasers and laser-like devices: part one. Australas J Dermatol. 2013 Aug;54(3):173-83. doi: 10.1111/ajd.12034. Epub 2013 Apr 10. PMID 23573909
- [Background] de Freitas LF, Hamblin MR. Proposed Mechanisms of Photobiomodulation or Low-Level Light Therapy. IEEE J Sel Top Quantum Electron. 2016 May-Jun;22(3):7000417. doi: 10.1109/JSTQE.2016.2561201. PMID 28070154
- [Background] Karu T. Mitochondrial mechanisms of photobiomodulation in context of new data about multiple roles of ATP. Photomed Laser Surg. 2010 Apr;28(2):159-60. doi: 10.1089/pho.2010.2789. No abstract available. PMID 20374017
- [Background] Clijsen R, Brunner A, Barbero M, Clarys P, Taeymans J. Effects of low-level laser therapy on pain in patients with musculoskeletal disorders: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2017 Aug;53(4):603-610. doi: 10.23736/S1973-9087.17.04432-X. Epub 2017 Jan 30. PMID 28145397
- [Background] Song HJ, Seo HJ, Kim D. Effectiveness of high-intensity laser therapy in the management of patients with knee osteoarthritis: A systematic review and meta-analysis of randomized controlled trials. J Back Musculoskelet Rehabil. 2020;33(6):875-884. doi: 10.3233/BMR-191738. PMID 32831189
- [Background] Song HJ, Seo HJ, Lee Y, Kim SK. Effectiveness of high-intensity laser therapy in the treatment of musculoskeletal disorders: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Dec;97(51):e13126. doi: 10.1097/MD.0000000000013126. PMID 30572425
- [Background] ElMeligie MM, Gbreel MI, Yehia RM, Hanafy AF. Clinical Efficacy of High-Intensity Laser Therapy on Lateral Epicondylitis Patients: A Systematic Review and Meta-analysis. Am J Phys Med Rehabil. 2023 Jan 1;102(1):64-70. doi: 10.1097/PHM.0000000000002039. Epub 2022 Apr 29. PMID 35512124
- [Background] Venosa M, Romanini E, Padua R, Cerciello S. Comparison of high-intensity laser therapy and combination of ultrasound treatment and transcutaneous nerve stimulation in patients with cervical spondylosis: a randomized controlled trial. Lasers Med Sci. 2019 Jul;34(5):947-953. doi: 10.1007/s10103-018-2682-7. Epub 2018 Nov 15. PMID 30443883
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Rampazo EP, de Andrade ALM, da Silva VR, Back CGN, Liebano RE. Photobiomodulation therapy and transcutaneous electrical nerve stimulation on chronic neck pain patients: Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Feb;99(8):e19191. doi: 10.1097/MD.0000000000019191. PMID 32080103
- [Background] Lim CY, In J. Randomization in clinical studies. Korean J Anesthesiol. 2019 Jun;72(3):221-232. doi: 10.4097/kja.19049. Epub 2019 Apr 1. PMID 30929415
- [Background] Ylinen J, Kautiainen H, Wiren K, Hakkinen A. Stretching exercises vs manual therapy in treatment of chronic neck pain: a randomized, controlled cross-over trial. J Rehabil Med. 2007 Mar;39(2):126-32. doi: 10.2340/16501977-0015. PMID 17351694
- [Background] Tunwattanapong P, Kongkasuwan R, Kuptniratsaikul V. The effectiveness of a neck and shoulder stretching exercise program among office workers with neck pain: a randomized controlled trial. Clin Rehabil. 2016 Jan;30(1):64-72. doi: 10.1177/0269215515575747. Epub 2015 Mar 16. PMID 25780258
- [Background] Sullivan GM, Feinn R. Using Effect Size-or Why the P Value Is Not Enough. J Grad Med Educ. 2012 Sep;4(3):279-82. doi: 10.4300/JGME-D-12-00156.1. No abstract available. PMID 23997866
- [Background] Kenareh R, Mirmohammadi SJ, Khatibi A, Shamsi F, Mehrparvar AH. The Comparison of The Efficacy of Photobiomodulation and Ultrasound in the Treatment of Chronic Non-specific Neck Pain: A Randomized Single-Blind Controlled Trial. J Lasers Med Sci. 2021 May 17;12:e20. doi: 10.34172/jlms.2021.20. eCollection 2021. PMID 34733743
- [Background] Modarresi S, Lukacs MJ, Ghodrati M, Salim S, MacDermid JC, Walton DM; CATWAD Consortium Group. A Systematic Review and Synthesis of Psychometric Properties of the Numeric Pain Rating Scale and the Visual Analog Scale for Use in People With Neck Pain. Clin J Pain. 2021 Oct 26;38(2):132-148. doi: 10.1097/AJP.0000000000000999. PMID 34699406
- [Background] Williams MA, McCarthy CJ, Chorti A, Cooke MW, Gates S. A systematic review of reliability and validity studies of methods for measuring active and passive cervical range of motion. J Manipulative Physiol Ther. 2010 Feb;33(2):138-55. doi: 10.1016/j.jmpt.2009.12.009. PMID 20170780
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Kubas C, Chen YW, Echeverri S, McCann SL, Denhoed MJ, Walker CJ, Kennedy CN, Reid WD. Reliability and Validity of Cervical Range of Motion and Muscle Strength Testing. J Strength Cond Res. 2017 Apr;31(4):1087-1096. doi: 10.1519/JSC.0000000000001578. PMID 27467513
- [Background] Andrade Ortega JA, Delgado Martinez AD, Almecija Ruiz R. Validation of the Spanish version of the Neck Disability Index. Spine (Phila Pa 1976). 2010 Feb 15;35(4):E114-8. doi: 10.1097/BRS.0b013e3181afea5d. PMID 20110848
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Background] Knapstad MK, Nordahl SHG, Naterstad IF, Ask T, Skouen JS, Goplen FK. Measuring pressure pain threshold in the cervical region of dizzy patients-The reliability of a pressure algometer. Physiother Res Int. 2018 Oct;23(4):e1736. doi: 10.1002/pri.1736. Epub 2018 Aug 7. PMID 30088327
- [Background] Waller R, Straker L, O'Sullivan P, Sterling M, Smith A. Reliability of pressure pain threshold testing in healthy pain free young adults. Scand J Pain. 2015 Oct 1;9(1):38-41. doi: 10.1016/j.sjpain.2015.05.004. PMID 29911647
- [Background] Rampazo da Silva EP, Silva VR, Bernardes AS, Matuzawa F, Liebano RE. Segmental and extrasegmental hypoalgesic effects of low-frequency pulsed current and modulated kilohertz-frequency currents in healthy subjects: randomized clinical trial. Physiother Theory Pract. 2021 Aug;37(8):916-925. doi: 10.1080/09593985.2019.1650857. Epub 2019 Aug 12. PMID 31402740
- [Background] Dundar U, Turkmen U, Toktas H, Solak O, Ulasli AM. Effect of high-intensity laser therapy in the management of myofascial pain syndrome of the trapezius: a double-blind, placebo-controlled study. Lasers Med Sci. 2015 Jan;30(1):325-32. doi: 10.1007/s10103-014-1671-8. Epub 2014 Oct 2. PMID 25274197
- [Derived] de la Barra Ortiz HA, Avila MA, Miranda LG, Liebano RE. Effect of high-intensity laser therapy in patients with non-specific chronic neck pain: study protocol for a randomized controlled trial. Trials. 2023 Aug 31;24(1):563. doi: 10.1186/s13063-023-07599-0. PMID 37653525